CLINICAL TRIAL: NCT03416868
Title: Preliminary Study 2 to Test the Effects of Ambulatory Voice Biofeedback in Small Groups of Patients With Vocal Hyperfunction
Brief Title: Preliminary Study 2 to Test the Effects of Ambulatory Voice Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Robert E Hillman, Research Director at the MGH Voice Center, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002849B; 1P50DC015446-01A1 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Vocal Fold Nodules; Muscle Tension Dysphonia
Keywords: Ambulatory; Biofeedback; Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care voice therapy with ambulatory voice biofeedback. (Experimental): Patients with Vocal Hyperfunction will undergo standard of care voice therapy, Ambulatory monitoring will be completed by the patients before therapy and throughout the first 3 weeks of therapy. Specifically, ambulatory monitoring will be worn by the patient for their 4 days with the most voicing during the first 3 weeks of therapy. Biofeedback will be activated only after the 2nd voice therapy session.
  Interventions: Behavioral: Ambulatory voice biofeedback

INTERVENTIONS:
Behavioral: Ambulatory voice biofeedback — Patients will be provided cues regarding their vocal behavior in daily life. Specifically, the patient will receive 100% feedback = a vibrotactile cue on a smartwatch every time the patient voices incorrectly. The specific objective voice measure for biofeedback will depend upon which measure is most strongly associated with improvements during voice therapy.

SUMMARY:
Patients with vocal hyperfunction will undergo standard of care voice therapy with ambulatory voice monitoring before therapy and after the first 3 voice therapy sessions. Biofeedback will be added to ambulatory monitoring after the 2nd voice therapy session only.

DETAILED DESCRIPTION:
This study will use a single subject design to determine if adding ambulatory voice biofeedback to conventional voice therapy can result in faster carryover (generalization) of new vocal behaviors established during voice therapy to daily life. Here, ambulatory voice biofeedback will be based on objective measures that have subject-specific sensitivity to vocal hyperfunction. Hypothesis: The ambulatory voice biofeedback week (week 2) will result in higher generalization percentages when compared to baseline and the week prior to the initiation of biofeedback (week 1). This effect will be retained when the biofeedback is removed (week 3), thus it will be different than baseline and week 1, but not different than week 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vocal fold nodules or muscle tension dysphonia undergoing voice therapy

Exclusion Criteria:

* If a patient's baseline ambulatory monitoring data is not at least 1 standard deviation away from a normative database in any measure, he/she will be excluded. Non-English speakers are excluded because prompts on the smartphone app are only available in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Hillman, PhD, Principal Investigator — Mass General Hospital, Harvard, MGH IHP
Locations (1):
- Massachusetts General Hospital - Center for Laryngeal Surgery and Voice Rehabilitation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Voice Therapy With Ambulatory Voice Biofeedback.
Started | 39
Completed | 36
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: There is a discrepancy in the numbers of enrolled patients here (total = 7) and compared to total enrolled (total = 39). This is because the first 32 patients' data were used to refine and adapt study protocols. The final 7 patients were acquired with this final protocol.
Arm/Group | Standard of Care Voice Therapy With Ambulatory Voice Biofeedback.
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 35 [18 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Percent compliance [Mean (Full Range); unit: Percentage of voicing below threshold] — Percentage compliance is the amount of voiced time patients spent below their biofeedback threshold divided by the total amount of voiced time. Each patient's biofeedback threshold was individually established with a voice measure associated with improved voicing during therapy.
  Percentage of voicing below threshold | 89.46 [78.23 to 98.67]

OUTCOME MEASURES:

1. Primary Outcome: Percent Compliance
Description: Using a patient-specific voice measure, patients will be asked to avoid crossing numeric thresholds. The amount of voicing spent within desired thresholds will be the "percent compliance".
Time Frame: Week 1, Week 2, Week 3
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: percentage of voicing crossing threshold
Groups:
- Standard of Care Voice Therapy With Ambulatory Voice Biofeedback.: Patients with Vocal Hyperfunction will undergo standard of care voice therapy. Ambulatory monitoring will be completed by the patients before therapy and throughout the first 3 weeks of therapy. Specifically, ambulatory monitoring will be worn by the patient for their 4 days with the most voicing during the first 3 weeks of therapy. Biofeedback will be activated only after the 2nd voice therapy session.
  Ambulatory voice biofeedback: Patients will be provided cues regarding their vocal behavior in daily life. Specifically, the patient will receive 100% feedback = a vibrotactile cue on a smartwatch every time the patient voices incorrectly. The specific objective voice measure for biofeedback will depend upon which measure is most strongly associated with improvements during voice therapy.
Arm/Group | Standard of Care Voice Therapy With Ambulatory Voice Biofeedback.
Number analyzed (Participants) | 7
percentage of voicing crossing threshold
  Week 1 | 89.04 [73.09 to 99.76]
  Week 2 | 92.44 [84.7 to 99.08]
  Week 3 | 90.76 [71.97 to 99.62]

ADVERSE EVENTS:
Time Frame: Patients were involved in this study for 3 weeks and adverse event data (anterior neck skin irritation) were collected at the end of each week.
Description: This is a low-risk clinical trial, as determined by the IRB. We will collect data only on Other Adverse Events, specifically patient-reported skin irritation where the monitor's sensor was taped to the neck during wear. Specifically, each patient will be systematically assessed for skin irritation by the investigator asking the patient if any skin irritation occurred at the end of each week of monitoring.
Arm/Group | Standard of Care Voice Therapy With Ambulatory Voice Biofeedback.
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03416868/Prot_SAP_ICF_000.pdf